CLINICAL TRIAL: NCT00203450
Title: Zonegran for the Treatment of Weight Gain Associated With Psychotropic Medication Use: A Placebo-Controlled Trial
Acronym: Zonegran
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Lori Davis, MD, ACOS R&D, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREAC Zonegran for Weight Loss; TREAC Zonegran for Weight Loss
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: obesity; zonisamide; zonegran; psychotropic weight gain; psychotropic
MeSH Terms: conditions — Obesity | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonegran (Experimental): Zonegran
  Interventions: Drug: Zonegran
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonegran — zonisamide
  Other Names: zonisamide
  Arms: Zonegran
Drug: Placebo — Placebo pill
  Other Names: placebo pill
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the efficacy of zonisamide (Zonegran; 100mg - 400mg/day) and placebo as an adjunctive agent on lowering weight in subjects who have a body mass index (BMI) of >25 and are on a psychotropic medication with a known side effect of weight gain.

DETAILED DESCRIPTION:
After the screening period, patients fulfilling entrance criteria will be randomized to 100mg of zonisamide or placebo in a 2:1 ratio respectively. Patients will be assessed at baseline and on Weeks 2, 4, 8, 12, and 16-post randomization for weight, side effects, and symptoms. Symptoms will be assessed by the Young Mania Rating Scale (YMRS), Brief Psychiatric Rating Scale (BPRS), Hamilton Depression Rating Scale (HAMD), Hamilton Rating Scale for Anxiety (HARS), and Self-report measures of general health and mental status at baseline, weeks 2, 4, 8, 12,and 16. At the conclusion of the study, patients will be tapered from the study medication and will return to their primary provider for continued treatment of their psychiatric condition.

ELIGIBILITY:
Inclusion Criteria:

* Are men or women, between the ages of 19 and 65, inclusive
* Have a diagnosis of any type of bipolar disorder or any type of psychotic disorder based on structured diagnostic interview (MINI).
* Are currently outpatients or inpatients and taking a neuroleptic or mood stabilizer medication (listed below) for the past 6 months, and on a stable dose for the past 2 months.
* Have a body mass index > 25.
* No substance use disorder in the past 2 months (except for nicotine or caffeine).
* Agree to not become pregnant during the study and agree to use an adequate method of birth control during the study such as a barrier method, hormonal contraceptive, or surgical sterilization (females only). All women of childbearing potential must have a negative pregnancy test before beginning study medication.
* Are able to swallow the capsules whole
* Are willing and able to follow Investigator instructions and study procedures, and report adverse events
* Not currently actively suicidal or homicidal.
* No use of topiramate within the last 6 months.
* No medical contraindication to the use of zonisamide.

List of medications for inclusion criterion #3:

All conventional neuroleptics. All atypical neuroleptics except aripiprazole or ziprasidone. All forms of valproate. All forms of lithium. All forms of carbamazepine.

Exclusion Criteria:

* Clinically significant renal or hepatic disease.
* History of acute intermittent porphyria, glucose-6phosphate dehydrogenase deficiency or hemolytic anemia.
* Allergy to zonisamide or sulfonamides.
* Have clinically unstable cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine, or other systemic disease
* Have laboratory test results that, in the opinion of the Investigator, are clinically significant abnormalities
* Require treatment with any medication (e.g., carbonic anhydrase inhibitors) that might interact adversely with, or obscure, the action of the study drug
* Are pregnant or lactating (females only)
* Have a history of nephrolithiasis
* Refuse to give informed consent
* Have previously enrolled in this study or previously been treated with zonisamide

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-05; Primary Completion 2005-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the efficacy of zonisamide (Zonegran; 100mg - 400mg/day) and placebo as an adjunctive agent on lowering weight in subjects who have a body mass index (BMI) of >25 and are on a psychotropic medication with

SECONDARY OUTCOMES:
NThe weight loss in patients treated with Zonisamide will be significantly greater than those treated with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research & Education Advancement Corporation, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Appolinario JC, Bueno JR, Coutinho W. Psychotropic drugs in the treatment of obesity: what promise? CNS Drugs. 2004;18(10):629-51. doi: 10.2165/00023210-200418100-00002. PMID 15270593